CLINICAL TRIAL: NCT04526782
Title: A Phase II Study of the BRAF Inhibitor Encorafenib in Combination With the MEK Inhibitor Binimetinib in Patients With BRAFV600E-mutant Metastatic Non-small Cell Lung Cancer
Brief Title: ENCOrafenib With Binimetinib in bRAF NSCLC
Acronym: ENCO-BRAF
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IFCT-1904
Record Dates: First submitted 2020-08-21; First posted 2020-08-26 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Non Small Cell Lung Cancer; BRAF V600E
Keywords: encorafenib; binimetinib; NSCLC; IFCT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — encorafenib; binimetinib

STUDY DESIGN:
Intervention Model Description: This is an open-label, multicenter, multi-cohort Phase 2 study of the combination of encorafenib and binimetinib in patients with previously treated and untreated BRAFV600E-mutant NSCLC.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (1st line) (Experimental): Encorafenib: 450 mg (6 × 75 mg capsule) QD Binimetinib: 45 mg (3 × 15 mg tablet) BID
  Interventions: Drug: Encorafenib 75 MG; Drug: Binimetinib 15 MG
- Cohort 2 (2nd line) (Experimental): Encorafenib: 450 mg (6 × 75 mg capsule) QD Binimetinib: 45 mg (3 × 15 mg tablet) BID
  Interventions: Drug: Encorafenib 75 MG; Drug: Binimetinib 15 MG

INTERVENTIONS:
Drug: Encorafenib 75 MG — 450 mg (6 × 75 mg capsule) per day
Drug: Binimetinib 15 MG — 45 mg (3 × 15 mg tablet) twice daily

SUMMARY:
A Phase II study of the BRAF inhibitor Encorafenib in combination with the MEK inhibitor Binimetinib in Patients with BRAFV600E-mutant metastatic Non-small Cell Lung Cancer

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have signed and dated an IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal subject care.

   Subjects must be willing and able to comply with scheduled visits, treatment schedule, and laboratory testing.
2. Male or female aged at least 18 years old.
3. Histologically confirmed diagnosis of NSCLC that is currently Stage IV (M1a, M1b or M1c AJCC 8th edition).
4. ECOG performance status of 0-1.
5. Able to swallow and retain oral medication.
6. Presence of a BRAFV600E mutation in lung cancer tissue as determined by a local laboratory assay.
7. The Investigator must confirm prior to enrolment that the patient has adequate tumor tissue available to determine BRAFV600E mutation status by central laboratory for confirmation.

   Note: Tumor tissue collected after the patient was diagnosed with metastatic disease is preferred.

   Tumor tissue sample must not be from locations previously radiated. Tumor sample must be 1 block or 10 to 15 unstained slides of analyzable tissue and one H&E slide.
8. Patients i) (COHORT A) who are either treatment-naïve (e.g., no prior systemic therapy for advanced/metastatic disease), ii) (COHORT B) who are in progression after having received 1) first-line platinum-based chemotherapy OR 2) first-line treatment with an anti-PD-1/L-1 inhibitor given alone or in combination with platinum-based chemotherapy or in combination with immunotherapy (e.g, ipilimumab) with or without platinum-based chemotherapy.

   Note: Alternative chemotherapy regimens are acceptable if the patient was platinum intolerant or ineligible.

   Patients with early stage disease (e.g., Stages I-III) who have had surgery followed by chemotherapy (e.g., treatment in the adjuvant setting), and present with new lesions or evidence of disease recurrence (e.g., metastatic disease), within 12 months of completing chemotherapy, would be considered as had received a first-line therapy.

   Maintenance therapy given after first-line therapy in the metastatic setting will not be considered a separate regimen, provided there was no documentation of disease progression between completion of first-line therapy and the start of maintenance therapy.
9. Presence of measurable disease based on RECIST v1.1.
10. Adequate bone marrow function characterized by the following at screening:

    i) ANC ≥ 1.5 × 109/L; ii) Platelets ≥ 100 × 109/L; iii) Hemoglobin ≥ 8.5 g/dL (with or without blood transfusions).
11. Adequate hepatic and renal function characterized by the following at screening:

    i) Total bilirubin ≤ 1.5 × ULN and < 2 mg/dL; OR total bilirubin >1.5 × ULN with indirect bilirubin < 1.5 × ULN; ii) ALT and AST ≤ 2.5 × ULN, or ≤ 5 × ULN in presence of liver metastases; iii) Serum creatinine ≤ 1.5 × ULN; or calculated creatinine clearance ≥ 50 mL/min by Cockcroft-Gault formula; or estimated glomerular filtration rate>50 mL/min/1.73m2.
12. Female patients of childbearing potential as described in Appendix 1, must have a negative serum β HCG test result.
13. Female patients of childbearing potential must agree to use methods of contraception that are highly effective or acceptable, as described in Appendix 1, and to not donate ova from Screening until 30 days after the last dose of study treatment.
14. Male patients must agree to use methods of contraception that are highly effective or acceptable, as described in Appendix 1, and to not donate sperm from Screening until 90 days after the last dose of encorafenib and binimetinib.
15. Patient covered by a national health insurance

Exclusion Criteria:

1. Patients with nonsquamous carcinoma who have documentation of any of the following: EGFR mutation, ALK fusion oncogene or ROS1 rearrangement.
2. Previous treatment with any other BRAF inhibitor (e.g., dabrafenib, vemurafenib…), or any other MEK inhibitor (e.g., trametinib, cobimetinib…) prior to screening and enrolment.

4. Patients who have received more than 1 prior line of systemic therapy in the advanced/metastatic setting for Cohort B.

Note: Generally, treatments that are separated by an event of progression are considered to represent another line of therapy.

Any therapeutic intervention including systemic therapy, surgery concurrent with or followed by systemic therapy, radiation concurrent with systemic therapy, or stereotactic radiation/radiosurgery, initiated or added to an existing therapy for oligometastatic disease will be considered a new line of therapy.

Palliative radiation to solitary lesions is permitted and will not be considered a new line of therapy.

Surgery/radiosurgery for CNS metastases is permitted and will not be considered a line of therapy as long as the surgery/radiosurgery was not given with systemic therapy (neoadjuvant or adjuvant).

Surgery followed by chemotherapy in the metastatic setting will be considered a line of therapy.

5. Receipt of anticancer therapies or investigational drugs within the following intervals before the first administration of study treatment: i) ≤14 days for chemotherapy, targeted small molecule therapy, radiation therapy, immunotherapy, or antineoplastic biologic therapy (e.g., erlotinib, crizotinib, bevacizumab etc.).

ii) ≤14 days or 5 half-lives (minimum of 14 days) for investigational agents or devices. For investigational agents with long half-lives (e.g., > 5 days), enrolment before the fifth half-life requires sponsor approval.

iii) Palliative radiation therapy must be complete 7 days prior to the first dose of study treatment.

6. Patients who have had major surgery (e.g., inpatient procedure with regional or general anesthesia) ≤ 6 weeks prior to start of study treatment.

7. For cohort B : Patient has not recovered to ≤Grade 1 from toxic effects of prior therapy and/or complications from prior surgical intervention before starting study treatment.

Note: Stable chronic conditions (≤ Grade 2) that are not expected to resolve (e.g., neuropathy, myalgia, alopecia, and prior therapy-related endocrinopathies) are exceptions.

8. Current use of a prohibited medication (including herbal medications, supplements, or foods), or use of a prohibited medication ≤1 week prior to the start of study treatment.

9. Impairment of gastrointestinal function or disease which may significantly alter the absorption of oral study treatment (e.g., uncontrolled nausea, vomiting or diarrhea, malabsorption syndrome, small bowel resection).

10. Impaired cardiovascular function or clinically significant cardiovascular diseases, including any of the following: i) History of acute myocardial infarction, acute coronary syndromes (including unstable angina, coronary artery bypass graft, coronary angioplasty or stenting) ≤ 6 months prior to start of study treatment; ii) Congestive heart failure requiring treatment (New York Heart Association Grade ≥2); iii) LVEF < 50% as determined by MUGA or ECHO; iv) Uncontrolled hypertension defined as persistent systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100 mmHg despite optimal therapy; v) History or presence of clinically significant cardiac arrhythmias (including uncontrolled atrial fibrillation or uncontrolled paroxysmal supraventricular tachycardia); vi) Baseline QTcF interval ≥480 ms or a history of prolonged QT syndrome. 11. History of thromboembolic or cerebrovascular events ≤12 weeks prior to the first dose of study treatment. Examples include transient ischemic attacks, cerebrovascular accidents, hemodynamically significant (i.e. massive or sub-massive) deep vein thrombosis or pulmonary emboli. Note: Patients with either deep vein thrombosis or pulmonary emboli that does not result in hemodynamic instability are allowed to enrol as long as they are on a stable dose of anticoagulants for at least 4 weeks. Note: Patients with thromboembolic events related to indwelling catheters or other procedures may be enrolled.

12. History or current evidence of RVO (Retinal Vein Occlusion) or current risk factors for RVO (e.g., uncontrolled glaucoma or ocular hypertension, history of hyper viscosity or hypercoagulability syndromes); history of retinal degenerative disease.

13. Concurrent neuromuscular disorder that is associated with the potential of elevated CK (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy).

14. Evidence of active, noninfectious pneumonitis, history of interstitial lung disease that required oral or intravenous glucocorticoid steroids for management.

15. Evidence of HBV or HCV infection. Note: Patients with laboratory evidence of cleared HBV or HCV infection may be enrolled. Note: Patients with no prior history of HBV infection who have been vaccinated against HBV and who have a positive antibody against hepatitis B surface antigen as the only evidence of prior exposure may enrol.

16. Patient who aas has a known history of a positive test for HIV or known AIDS.

17. Active infection requiring systemic therapy. 18. Patients with symptomatic brain metastasis, leptomeningeal disease or other active CNS metastases are not eligible.

Note: Patients with previously treated or not treated brain metastases may participate provided they are stable (e.g., without evidence of progression by radiographic imaging for at least 28 days before the first dose of study treatment and neurologic symptoms have returned to baseline) Patients must have no evidence of new or enlarging brain metastases or CNS edema.

Patient must have discontinued use of steroids at least 7 days before the first dose of study treatment.

19. Concurrent or previous other malignancy within 2 years of study entry, except curatively treated basal or squamous cell skin cancer, prostate intraepithelial neoplasm, carcinoma in-situ of the cervix, Bowen's disease and Gleason 6 prostate cancer.

20. Known sensitivity or contraindication to any component of study treatment or their excipients.

21. Pregnancy confirmed by a positive β-HCG laboratory test result, or breastfeeding (lactating).

22. Other severe, acute or chronic medical or psychiatric condition(s) or laboratory abnormality that may increase the risk associated with study participation or study treatment administration or that may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient an inappropriate candidate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Estimated)
Dates: Start 2021-01-19 (Actual); Primary Completion 2025-07-16 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 6 months
  Objective Response Rate at 6 months using RECIST1.1 criteria

SECONDARY OUTCOMES:
Duration Response Rate | about 12 months
  Time from the date of the first documented response (CR or PR) to the earliest date of disease progression (RECIST 1.1), or death due to any cause.
Progression-free Survival | about 24 months
  Time from enrollment to first observation of progression (RECIST1.1) or date of death (from any cause)
Overall Survival | about 24 months
  Time from enrollment until death due to any cause
Incidence, type and severity of adverse events | From time of informed consent through treatment period and up to 30 days post last dose of study treatment (about 24 months)
  Descriptive statistics of safety will be presented using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: David Planchard, Principal Investigator — Gustave Roussy (Villejuif - France); Charles Ricordel, Principal Investigator — CHU Rennes,France
Locations (36):
- France (36):
  - Annemasse - CH, Ambilly
  - Angers - CHU, Angers
  - Avignon - Institut Sainte-Catherine, Avignon
  - Bordeaux - Institut Bergonié, Bordeaux
  - Boulogne - Ambroise Paré, Boulogne-Billancourt
  - Brest - CHU, Brest
  - Caen - CHU Côte de Nacre, Caen
  - CH, Colmar
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Centre Georges François Leclerc, Dijon
  - CHRU Grenoble, Grenoble
  - La Roche Sur Yon - CH, La Roche-sur-Yon
  - CH Le Mans, Le Mans
  - CHRU de Lille, Lille
  - CHU Dupuytren, Limoges
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - AP-HM Hôpital Nord, Marseille
  - Montpellier - CHRU, Montpellier
  - Mulhouse - GHRMSA, Mulhouse
  - Nancy - Institut de Cancérologie de Lorraine, Nancy
  - Centre Antoine LACASSAGNE, Nice
  - AP-HP Hôpital Cochin, Paris
  - AP-HP Hôpital Tenon, Paris
  - Hôpital BICHAT, Paris
  - Paris - Institut Curie, Paris
  - Centre Hospitalier Général - Pau, Pau
  - Lyon - URCOT, Pierre-Bénite
  - CHU Rennes - Hôpital Pontchaillou, Rennes
  - CHU Charles Nicolle, Rouen
  - Saint Quentin - CH, Saint-Quentin
  - Nouvel Hôpital Civil - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - CHU Toulouse - Pneumologie, Toulouse
  - Tours - CHU, Tours
  - Villefranche-Sur-Saône - Hôpital Nord-Ouest, Villefranche-sur-Saône
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data underlying the results reported in this article, as well as the study protocol and statistical analysis plan, will be made available after deidentification immediately following publication and for three years. Researchers who provide a methodologically sound proposal for any purpose may direct proposals to contact@ifct.fr. To gain access, data requestors will need to sign a data access agreement that requires approval by the French Cooperative Thoracic Intergroup.

REFERENCES:
- See also: IFCT website — https://www.ifct.fr/etudes-cliniques/139-ifct-1904